CLINICAL TRIAL: NCT04125017
Title: Comparative Study Between Two Techniques for Artificial Shrinkage of Blastocysts Prior to Vitrification: LASER Pulse Versus Micro-needle Technique in Increasing Chemical, Clinical Pregnancy and Live Birth Rates After ICSI
Brief Title: Atrificial Shrinkage of Blastocyst Before In Vitro Fertilization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aljazeera Hospital (Other)
Collaborators: Adam International Hospital (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Consultant of Obstetrics and Gynecology, Aljazeera Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: blastocyst preparation
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Intervention Model Description: effect of using LASER pulse versus micro-needle use in the artificial shrinkage of blastocysts .
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- effect of using LASER pulse (Other): effect of using LASER pulse versus micro-needle use in the artificial shrinkage of blastocysts as a previous step before vitrification in regarding their effect on embryo viability
  Interventions: Device: ICSI with laser pulse; Device: ICSI with micro needle technique
- Micro-needle Technique (Other): effect of using LASER pulse versus micro-needle use in the artificial shrinkage of blastocysts as a previous step before vitrification in regarding their effect on embryo viability
  Interventions: Device: ICSI with laser pulse; Device: ICSI with micro needle technique

INTERVENTIONS:
Device: ICSI with laser pulse — Using laser pulse before ICSI
Device: ICSI with micro needle technique — Using micro needle technique before ICSI

SUMMARY:
Vitrification is a modern cryopreservation technique based on sudden cooling of reproductive cells to a temperature of -196 ° C in seconds that produces glass-like solidification of a solution without crystallization, but by extreme elevation in viscosity during freezing

DETAILED DESCRIPTION:
Vitrification is a modern cryopreservation technique based on sudden cooling of reproductive cells to a temperature of -196 ° C in seconds that produces glass-like solidification of a solution without crystallization, but by extreme elevation in viscosity during freezing Unlike the slow freezing method, vitrification has better results in a complete elimination of ice crystal inside the cells as well as in the surrounding solution -Also, it has a significantly higher post-thawing survival rate in comparison to slow freezing method

ELIGIBILITY:
Inclusion Criteria:

* women with infertility from 20 to 44 years

Exclusion Criteria:

* women with age more than 44 or less than 20

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Females who have infertility
Enrollment: 409 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-02-05 (Actual)

PRIMARY OUTCOMES:
The number of women who will have positive pregnancy test | 2 months
  The number of women who will come pregnant after each technique

CONTACTS AND LOCATIONS:
Overall Officials: manal kamel, Principal Investigator — Adam hospital
Locations (1):
- Adam, Giza, Egypt

REFERENCES:
- [Derived] Kamel Mohamed M, El-Noury MAH, Amer MK, Fakhry E, Alalfy M. Comparative study between two techniques for artificial shrinkage of blastocysts prior to vitrification: LASER pulse versus micro-needle technique in increasing chemical, clinical pregnancy and live birth rates after ICSI, a randomized controlled trial. J Matern Fetal Neonatal Med. 2022 Dec;35(25):4910-4917. doi: 10.1080/14767058.2021.1873265. Epub 2021 Feb 28. PMID 33645399